CLINICAL TRIAL: NCT00299455
Title: Phase 4 Efficacy Study of Antimicrobials in the Treatment of Acute Otitis Media in Young Children
Brief Title: Amoxicillin Clavulanate in Treatment of Acute Otitis Media
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Turku (Other)
Collaborators: Finnish Institute for Health and Welfare (Other Government)
Responsible Party: Aino Ruohola, Department of Pediatrcis, Turku University Hospital, Turku, Finland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RRR-60
Record Dates: First submitted 2006-03-03; First posted 2006-03-06 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Acute Otitis Media
MeSH Terms: conditions — Otitis Media | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Reconstituted amoxicillin-clavulanate at 40/5.7 mg/kg/day in 2 divided doses for 7 days.
  Interventions: Drug: amoxicillin-clavulanate
- 2 (Placebo Comparator): Reconstituted placebo in 2 divided doses for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: amoxicillin-clavulanate — Amoxicillin clavulanate 40 mg/kg/day divided into two daily doses for 7 days. Capsules will be produced by pulverizing amoxicillin clavulanate tablets (Augmentin 875 mg; manufacturer Glaxo SmithKline Beecham; ATC Code: J01CR02) and mixing that with lactose monohydrate. Each capsule will contain Augmentin tablet powder 68 mg and lactose monohydrate 572 mg. This means amoxicillin 40 mg and clavulanate 5,7 mg respecting the dose per 2 kg.
  Arms: 1
Drug: Placebo — Placebo twice a day for 7 days. Placebo capsules contain lactose monohydrate 640 mg.
  Arms: 2

SUMMARY:
This is a prospective, randomized, double-blind, placebo controlled one-center study carried out in primary care setting of the health center of City of Turku, Finland. The study patients will be allocated to one of the two parallel treatment groups (amoxicillin-clavulanate or placebo). The hypothesis is that the symptoms and signs of acute otitis media are resolved more effectively with antimicrobial treatment than with placebo. Furthermore, this study aims at finding out prognostic factors that could help to direct antimicrobial treatment for correct subgroups of young patients.

ELIGIBILITY:
Inclusion Criteria:

* Acute otitis media
* Age 6 - 35 mo

Exclusion Criteria:

* Spontaneous perforation of the tympanic membrane and drainage
* Systemic or nasal corticosteroid therapy within 3 preceding days
* Antihistamine therapy with 3 preceding days
* Oseltamivir therapy within 3 preceding days
* Allergy to amoxicillin/penicillin
* Tympanostomy tube present in tympanic membrane
* Clinical evidence of infection requiring systemic antimicrobial treatment
* Documented Ebstein Barr virus infection within 7 preceding days
* Down syndrome or other condition to affect middle ear infections
* Known immunodeficiency
* Vomiting or another symptom to violate per oral dosage
* Poor parental co-operation due to language or other reasons
* Use of any investigational drugs during the 4 preceding weeks

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2006-03; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Compare time to treatment failure in children receiving amoxicillin-clavulanate to children receiving placebo | During the first 8 days of follow-up

SECONDARY OUTCOMES:
Time to resolution of symptoms in children receiving amoxicillin-clavulanate to children receiving placebo | Duration of study
Time to resolution of acute inflammatory signs of middle ear | Duration of study
Compare the 2 treatment groups regarding the doses of analgesic medication and number of days analgesics are administered by children's parents | First 7 days of follow-up
Compare the 2 treatment groups regarding the number of days with absenteeism from day care and/or parental absenteeism from work | First 7 days of follow-up
Compare the incidence of adverse events accompanying the 2 treatment regimens | Duration of study
Time to resolution of middle ear fluid in the ear(s) that is affected on study day 1 | Duration of study
Time to relapse of acute otitis media | Study days 9-17
Time to first reinfection of acute otitis media | From study day 18 to the end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Aino Ruohola, MD, PhD, Principal Investigator — Pediatrician
Locations (2):
- Finland (2):
  - Department of Pediatrics, Turku University Hospital, Turku
  - Turku

REFERENCES:
- [Derived] Uitti JM, Salantera S, Laine MK, Tahtinen PA, Ruohola A. Adaptation of pain scales for parent observation: are pain scales and symptoms useful in detecting pain of young children with the suspicion of acute otitis media? BMC Pediatr. 2018 Dec 20;18(1):392. doi: 10.1186/s12887-018-1361-y. PMID 30572868
- [Derived] Ruohola A, Laine MK, Tahtinen PA. Effect of Antimicrobial Treatment on the Resolution of Middle-Ear Effusion After Acute Otitis Media. J Pediatric Infect Dis Soc. 2018 Feb 19;7(1):64-70. doi: 10.1093/jpids/pix008. PMID 28340091
- [Derived] Laine MK, Tahtinen PA, Ruuskanen O, Loyttyniemi E, Ruohola A. Can trained nurses exclude acute otitis media with tympanometry or acoustic reflectometry in symptomatic children? Scand J Prim Health Care. 2015;33(4):298-304. doi: 10.3109/02813432.2015.1118835. Epub 2015 Dec 14. PMID 26651157
- [Derived] Erkkola-Anttinen N, Laine MK, Tahtinen PA, Ruohola A. Parental role in the diagnostics of otitis media: can layman parents use spectral gradient acoustic reflectometry reliably? Int J Pediatr Otorhinolaryngol. 2015 Sep;79(9):1516-21. doi: 10.1016/j.ijporl.2015.06.040. Epub 2015 Jul 6. PMID 26183005
- [Derived] Tahtinen PA, Laine MK, Huovinen P, Jalava J, Ruuskanen O, Ruohola A. A placebo-controlled trial of antimicrobial treatment for acute otitis media. N Engl J Med. 2011 Jan 13;364(2):116-26. doi: 10.1056/NEJMoa1007174. PMID 21226577
- [Derived] Laine MK, Tahtinen PA, Ruuskanen O, Huovinen P, Ruohola A. Symptoms or symptom-based scores cannot predict acute otitis media at otitis-prone age. Pediatrics. 2010 May;125(5):e1154-61. doi: 10.1542/peds.2009-2689. Epub 2010 Apr 5. PMID 20368317